CLINICAL TRIAL: NCT06090682
Title: Effect and Mechanism of Deep Brain Stimulation and Transcranial Magnetic Stimulation on Parkinson's Disease With Cognitive Impairment
Brief Title: Effect and Mechanism of Brain Stimulation for Parkinson's Disease With Cognitive Impairment
Status: Recruiting | Type: Observational
Sponsor: Tianjin Huanhu Hospital (Other)
Responsible Party: Principal Investigator, Guangrui Zhao, Associate Professor, Tianjin Huanhu Hospital
Other Study IDs: TianjinHH-02
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease; Cognitive Impairment
Keywords: Parkinson Disease; Cognitive Impairment; Deep brain stimulation; Transcranial magnetic stimulation
MeSH Terms: conditions — Parkinson Disease; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cognitive Impairment (CI) group and No Cognitive Impairment (NCI) group: We intend to recruit 200 patients with primary PD to undergo DBS surgery or only TMS treatment according to whether the surgical indication is available. We will observe the changes in cognitive function of patients before and after different brain stimulation treatments.
  Parkinson's disease patients with cognitive impairment after brain stimulation were divided into cognitive impairment group, and those without cognitive impairment after treatment were divided into no cognitive impairment group
  Interventions: Device: Deep Brain Stimulation(DBS) and Transcranial Magnetic Stimulation(TMS)

INTERVENTIONS:
Device: Deep Brain Stimulation(DBS) and Transcranial Magnetic Stimulation(TMS) — We observed the changes in cognitive function of patients before and after different brain stimulation treatments, and further compared the effects of different brain stimulation treatments on cognitive function of PD patients and the related mechanisms according to whether DBS surgery was performed or TMS therapy was given only according to the surgical indications.

SUMMARY:
This study intends to apply structural and functional brain network neuroimaging techniques combined with image post-processing methods to explore the differences in brain network changes in PD patients with cognitive impairment after DBS or TMS.

DETAILED DESCRIPTION:
A variety of post-processing methods (VBM, SPM, CAT, LEAD-DBS, etc.) were used to analyze structural brain network images (sMRI, DTI) and functional brain network images (rs-fMRI, PET) based on connectomics, and combined with the changes of clinical symptoms before and after treatment. To study the mechanism of the influence of neural regulation on brain network, and further analyze how DBS and TMS improve the cognitive symptoms of PD patients from the perspective of brain connectomics, so as to explore the occurrence and development of Parkinson's disease with cognitive impairment and the possible improvement mechanism.According to the individual differences in clinical symptoms of different PD patients, better stimulation sites and the best brain network are sought to further guide the surgical plan, so as to obtain the best clinical treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. The clinical diagnosis of PD is consistent with the United Kingdom Parkinson's Disease Society Brain Bank criteria, with disease duration over 5 years, acute levodopa motor response ≥30%, and indication for STN-DBS.

Exclusion Criteria:

Exclusion criteria included patients with severe cognitive impairment, severe psychiatric disorders, acute levodopa motor response less than 30%, atypical parkinsonism, and contraindications to surgery.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Recruiting 200 patients with primary Parkinson's disease, aged less than 75 years old, regardless of gender, without prior brain injury, and with a history of brain surgery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Rating Scale(MoCA) | December 2023 to December 2026
  The Montreal Cognitive Rating Scale was used to assess the overall cognitive status of patients before and after treatment
verbal fluency test (VF) | December 2023 to December 2026
  VF test was used to assess frontal executive function and related language function

SECONDARY OUTCOMES:
the third part of the Unified Parkinson's Disease Rating Scale (UPDRS III) | December 2023 to December 2026
  Measures motor symptoms and Higher scores indicate more severe impairment in motor function

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
We observed the therapeutic effects of DBS and TMS on cognitive impairment in patients with Parkinson's disease and analyzed the possible mechanisms of cognitive changes